CLINICAL TRIAL: NCT02976363
Title: Study of Maximal Respiratory Pressures After Exposure to Breast Radiotherapy in Women
Brief Title: Maximal Respiratory Pressures After Radiotherapy
Status: Completed | Type: Observational
Sponsor: Federal University of Mato Grosso (Other)
Responsible Party: Principal Investigator, Thays Mello de Avila, Principal Investigator, Federal University of Mato Grosso
Other Study IDs: 46913415700000021
Record Dates: First submitted 2016-11-18; First posted 2016-11-29 (Estimated); Last update posted 2016-11-29 (Estimated); Status verified 2016-11

CONDITIONS: Respiratory Function Tests
Keywords: Radiotherapy; Respiratory muscles; Neoplasms; Breast
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Quadrantectomy Group: The Quadrantectomy Group sample performed adjuvant radiotherapy with a linear accelerator, whose the total dosage was 5000 centigray (cGy), the daily dose 200 cGy distributed into twenty-five sessions, totaling 25 days of treatment. And data from Maximal Respiratory Pressures (MIP/MEP) were collected at two phases in the sample of Quadrantectomy Group: before the first session of radiotherapy and after the twenty-fifth session corresponding to the last day of the radiotherapy treatment.
  Interventions: Radiation: Radiotherapy breast cancer; Other: Evaluation Maximal Respiratory Pressures
- Control Group: While for the control group women with no breast cancer history were invited. Data from Maximal Respiratory Pressures (MIP/MEP) were collected at one phase in the sample of control group.
  Interventions: Other: Evaluation Maximal Respiratory Pressures

INTERVENTIONS:
Radiation: Radiotherapy breast cancer
  Groups: Quadrantectomy Group
Other: Evaluation Maximal Respiratory Pressures
  Other Names: MIP and MEP

SUMMARY:
Objective: The purpose of this research was to study the Maximal Respiratory Pressures (MRP) after exposure to breast radiation therapy in women. Methods: Prospective observational study performed at the Hospital de cancer Alfred in Campo Grande/MS. The sample of this study consisted of women (N = 16) divided into two groups: women exposed to breast radiotherapy after underwent quadrantectomy surgery (n = 8); and women with no history of cancer (n = 8). We evaluated the strength of respiratory muscles through the Maximal Inspiratory Pressure (MIP) and Maximal Expiratory Pressure (MEP) using the handset called manovacuometer. The examination was performed before the first session and after the twenty-fifth session related to the last day of the radiation treatment; evaluation of anthropometric data of weight and height to detect the body mass index (BMI); evaluation of clinical respiratory symptoms of dyspnea using the Medical Research Council (MRC) Dyspnea Scale and characterization of cough with Common Pulmonary Toxicity Criteria, in the classification of clinical pneumonitis.

DETAILED DESCRIPTION:
Study design and sample The research consisted of an observational prospective study with control group. The study was approved by the Ethics Committee of the Federal University of Mato Grosso do Sul (UFMS) with the number 46913415.7.0000.002. All participants signed an informed consent form after being informed about the design and objectives of the study according to Resolution 466/12 of the National Council of Health Ministry of Health (CNS).

The quadrantectomy group participants were selected consecutively among patients who initiated radiotherapy. While the control group was selected during routine exams of he image sector from Hospital de Cancer Alfred Abrão.

Research site The execution of the research took place in the Radiotherapy sector of Hospital de Cancer Alfred Abrão in Campo Grande - Mato Grosso do Sul state, from December 2015 to February 2016.

Radiotherapy Protocol The Quadrantectomy Group sample performed adjuvant radiotherapy with a linear accelerator, whose the total dosage was 5000 centigray (cGy), the daily dose 200 cGy distributed into twenty-five sessions, totaling 25 days of treatment.

PROCEDURES Evaluation of maximal respiratory pressures (MRP) Quantification of MIP and MEP was performed with the portable device called manometer, Wika brand with pressure scale ranging from -150 to 150 centimeters of water (0 to -150 to (0 to -150 for MIP; 0 to 150 for MEP). The mouthpiece attached to the device had a hole of 2 mm in diameter, in order to function as a relief valve of the facial muscles. During the measurement of maximal respiratory pressures, the survey participants remained in seated position with the trunk in a 90 ° angle with the lower limbs. A forced expiration was requested until reaching the residual volume (RV) for the measurement of MIP, followed by a maximal inspiratory effort against the occluded airway (Maneuver Muller), this maneuver kept for up to 2 seconds. While the evaluation of MEP, a maximum inspiration was requested to Total Lung Capacity (TLC), followed by a maximal expiratory effort against the occluded airway (Muller maneuver), maintained for up to 2 seconds.

Data from Maximal Respiratory Pressures were collected at two phases in the sample of quadrantectomy group: before the first session of radiotherapy and after the twenty-fifth session corresponding to the last day of the radiotherapy treatment.

The evaluation of the MRP was performed according to the Brazilian Guidelines for Pulmonary Function Tests. The results were analyzed according to the predictive values of Neder regression equations (1999).

Complementary evaluation Anthropometric data evaluated to detect the body mass index (BMI) were: weight and height. Evaluation of dyspnea and cough symptoms with modified Dyspnea Medical Research Council scale (MRC) with the Common Pulmonary Toxicity Common Criteria scale (CTC Version 2.0) was performed to classify the clinic pneumonitis according to the Common Toxicity Criteria (CTC Version 2.0).

Statistics The variables classified as dependent were the maximal respiratory pressures. While the independent variables were sex, age, weight, height, BMI.

The comparison data analysis between the control group and quadrantectomy in relation to the variables: age, height, weight, BMI, MIP and MEP, was performed using the student's t test. The comparison between the moments before and after the radiotherapy in relation to MIP and MEP was performed using the student's t test paired, considering a 5% significance level. The other results of this study were presented in the form of descriptive statistics or in tables and graphics. Statistical analysis was performed using the sigma plot version 12.5 statistical program.

ELIGIBILITY:
Inclusion Criteria:

* There were selected women aged 40-70 years old, breast quadrantectomy post-surgery and adjuvant radiotherapy indication to compose the experimental group.
* While for the control group women aged 40-70 years old with no breast cancer history were invited.

Exclusion Criteria:

* The exclusion of the experimental and control groups were based on the following criteria:
* lung disease association, central or peripheral neurological disorders, refusal to participate in the study, difficulties in understanding and the completion of the protocol tests.
* The unique criteria of the experimental group were: metastatic cancer, concomitant chemotherapy to radiotherapy, hormone therapy and withdrawal of treatment.

Ages: 40 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The quadrantectomy group (QG) participants were selected consecutively among patients who initiated radiotherapy. While the control group (CG) was selected during routine exams of he image sector from Hospital de Cancer Alfred Abrão.
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2015-12; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Maximal Respiratory Pressures (MRP) after exposure to breast radiation therapy in women | three months

CONTACTS AND LOCATIONS:
Overall Officials: Thays M Avila, Principal Investigator — UFMS

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Black LF, Hyatt RE. Maximal respiratory pressures: normal values and relationship to age and sex. Am Rev Respir Dis. 1969 May;99(5):696-702. doi: 10.1164/arrd.1969.99.5.696. No abstract available. PMID 5772056
- [Background] Neder JA, Andreoni S, Lerario MC, Nery LE. Reference values for lung function tests. II. Maximal respiratory pressures and voluntary ventilation. Braz J Med Biol Res. 1999 Jun;32(6):719-27. doi: 10.1590/s0100-879x1999000600007. PMID 10412550
- [Background] Spyropoulou D, Leotsinidis M, Tsiamita M, Spiropoulos K, Kardamakis D. Pulmonary function testing in women with breast cancer treated with radiotherapy and chemotherapy. In Vivo. 2009 Sep-Oct;23(5):867-71. PMID 19779125
- [Background] Lee TF, Chao PJ, Chang L, Ting HM, Huang YJ. Developing Multivariable Normal Tissue Complication Probability Model to Predict the Incidence of Symptomatic Radiation Pneumonitis among Breast Cancer Patients. PLoS One. 2015 Jul 6;10(7):e0131736. doi: 10.1371/journal.pone.0131736. eCollection 2015. PMID 26147496